CLINICAL TRIAL: NCT03410212
Title: Efficacy of Ketorolac and Lidocaine Inferior Alveolar Nerve Blocks in Patients With With Symptomatic Irreversible Pulpitis: a Prospective Double Blind, Randomized Clinical Trial
Brief Title: Efficacy of Block Injection of an Anti Inflammatory Medicine in Patients With Mandibular Dental Pain
Acronym: IANB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nahid Mohammadzadeh Akhlaghi, Associate Professor, Azad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.IAU.DENTAL.REC.1396,31
Record Dates: First submitted 2018-01-04; First posted 2018-01-25 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Inferior alveolar nerve block; ketorolac; success
MeSH Terms: interventions — Ketorolac Tromethamine; Ketorolac; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac Tromethanine (Active Comparator): In the experimental group, 30mg/mL, ketorolac tromethamine will be injected as same as the first IANB and 5 minutes following it.
  Interventions: Drug: Ketorolac Tromethamine
- No injection (Sham Comparator): In the control group, 5 minutes following the IANB, the sham injection will be provided at the same place of the first injection.
  Interventions: Behavioral: Sham injection

INTERVENTIONS:
Drug: Ketorolac Tromethamine — The 30mg/mL vial of Ketorolac will be injected as second inferior alveolar nerve block and the success of anesthesia will be evaluated using visual analog scale.
  Other Names: Toradol, Acular, Sprix
  Arms: Ketorolac Tromethanine
Behavioral: Sham injection — In the control group, the sham injection will be provided at the same place of the first inferior alveolar nerve block but any injection would be done.
  Arms: No injection

SUMMARY:
The aim of this study is to determine whether inferior alveolar nerve block of ketorolac and lidocaine would improve the success rate in teeth with symptomatic irreversible Pulpitis.

Design: In this randomized double-blind clinical trial, sixty healthy adult volunteers with including criteria have been randomly divided into two groups (n=30). Following the 5 minutes of the first IANB using 1.8 ml 2% lidocaine 2% containing 1:100000, the patients of case group have received a standard inferior alveolar nerve block injection that used 1 ml ketorolac tromethamine 30 mg/ml. The patients of the control group received a sham injection. After achieving the lip numbness, access preparation initiated after 15 minutes of initial IANB with two negative responses to the electric pulp test. Any pain during caries and dentin removal, access cavity preparation, and root canal preparation have been recorded using analog visual scale (HP-VAS). The success was considered as none or mild pain during treatment. The data have been analyzed using Mann-U-Whitney test.

Intervention main outcome measures: Pain during caries and dentin removal access cavity preparation, and root canal preparation using VAS.

DETAILED DESCRIPTION:
The aim of this study is to determine whether inferior alveolar nerve block of ketorolac and lidocaine would improve the success rate in teeth with symptomatic irreversible Pulpitis. Design: In this randomized double-blind clinical trial, sixty healthy adult volunteers with including criteria have been randomly divided into two groups (n=30). All patients have been received standard inferior alveolar nerve block injection that used 1.8 ml 2% lidocaine 2% containing 1:100000 after negative aspiration. After 5 minutes 30 patients have received a standard inferior alveolar nerve block injection that used 1 ml ketorolac tromethamine 30 mg/ml. the other 30 patients received a sham injection. After achieving the lip numbness, the pulp anesthesia has been evaluated after 5 minutes by using electric pulp tester (Pakell Inc, Edgewood, NY). Endodontic access preparation initiated after 15 minutes of initial IANB with two negative responses to the electric pulp test. Any pain during caries and dentin removal, access cavity preparation, and root canal preparation have been recorded using analog visual scale (HP-VAS). The success was considered as none or mild pain during treatment. The data have been analyzed using Mann-U-Whitney test.Participants including major eligibility criteria: all patients with symptomatic irreversible pulpitis (HP VAS ≥54) of a mandibular molar tooth without systemic diseases; nonsmoking; without any medicine consumption or analgesic and sedation Intervention Main outcome measures: Pain during caries and dentin removal, access cavity preparation, and root canal preparation using VAS.

ELIGIBILITY:
Inclusion Criteria:

* patients with age ranged 18-65
* without systemic diseases;
* without any medicine consumption;
* nonsmoking;
* nonpregnant;
* non-breastfeeding;
* with symptomatic irreversible pulpitis (Visual Analog Scale ≥ 54) in one mandibular
* the molar that needs root canal treatment

Exclusion Criteria:

* patients under 18 or above 65 years old
* with systemic diseases;
* with any medicine consumption;
* smoking;
* pregnant;
* breastfeeding;
* without symptomatic irreversible pulpitis (Visual Analog Scale ≥ 54) in one mandibular
* the molar that needs root canal treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
pain during the root canal treatment | Average of 1 year
  Any pain during caries/dentin removal, access cavity and root canal preparation will be evaluated using 170 mm visual analog scale. Lack of pain or pain equal or less than 54 will be deemed success of anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Branch, AZad UMS, Tehran, Iran